CLINICAL TRIAL: NCT06073834
Title: LUNG INFECTION in ICU
Brief Title: LUNG INFECTION in ICU (LUNG-I3)
Acronym: LUNG-I3
Status: Recruiting | Type: Observational
Sponsor: BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: LUNG-I3
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: VAP - Ventilator Associated Pneumonia
Keywords: VAP - Ventilator Associated Pneumonia; Sepsis; Lung Infection; Broncho-alveolar Lavage; ICU
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Four types of samples are taken for the study per patient at day 4 after ICU admission:
  * whole blood collected in a PAXgene tube
  * dry tube for serum biobank
  * lithium heparin tube for plasma biobank
  * bronchoalveolar Lavage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
objective of LUNG-I3 study is to assess the quantitative and functional differences in cells between blood and bronchoalveolar lavage (BAL) fluid after an infection, with a special focus on alveolar macrophages and neutrophils

ELIGIBILITY:
Inclusion Criteria:

All the following criteria

* Age 18 years or greater
* Severe ICU patients hospitalized for one of the above diseases:

  * Septic shock (requirement of vasopressor to maintain a mean arterial pressure of 65 mm Hg or greater and serum lactate level greater than 2 mmol/L (>18 mg/dL) in the absence of hypovolemia) caused either by pneumonia (n=20) or another source n=20)
  * Severe trauma (level I and II), Injury Severity Score ≥ 25 OR
  * Burn with TBSA over 20%
* NAD > 0.1 µg/kg/min
* At least 2 SOFA criteria ≥ 2 points

Exclusion Criteria:

* Aspiration pneumonia
* Unable to obtain a valid and written consent from a patient or their legally authorized representative in accordance with the local regulatory instances (this includes in FR: Person not affiliated to a health insurance scheme, or not a beneficiary of such a scheme. Persons who are the subject of a legal protection order. Person with restricted freedom following a legal or administrative decision and a person admitted without their consent pursuant to Articles L.3212-1 and 3213-1, which are not included in Article L.1121-8 of the French Public Health Code.)
* COPD
* Smoke inhalation in burn patients
* Participation in an intervention study
* Pregnant or breastfeeding women
* Immunocompromised patients, defined as

  * patients with solid tumors with chemotherapy in the last 3 months or a progressive metastatic disease
  * hematologic malignancies
  * solid organ transplantation
  * HIV infection with or without AIDS
  * treatment with corticosteroids (> 3 months at any dosage or ≥ 1 mg/kg prednisone equivalent per day for > 7 day)
  * treatment with other immunosuppressive drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU Adult patients hospitalized and managed for septic shock or severe trauma (including severe burn) and undergoing mechanical ventilation (within 24h of admission) with an expected length upper than 3 days.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
immune cells patterns in VAP | before and at time of VAP diagnosis
  The primary endpoint will be to describe and compare the distribution of immune cells within the lung and the blood before VAP diagnosis (VAP prediction) and at the time of VAP diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Edouard Herriot, Lyon, France